CLINICAL TRIAL: NCT03477422
Title: Randomized, Double-blind, Double-dummy, Active-controlled, Multi-centre Trial to Compare the Efficacy and Safety of CSE-1034 (Ceftriaxone+ Sulbactam+ EDTA) With Meropenem in Infections Caused by β-Lactamase (ESBL and MBL) Producing Gram-Negative Bacteria
Brief Title: CSE-1034 (Ceftriaxone+ Sulbactam+ EDTA) Compared to Meropenem in Complicated Urinary Tract Infections (cUTIs) Caused by ESBL Producing Gram Negative Bacteria
Acronym: PLEA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Venus Remedies Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VRL/CSE-1034/05/2012; CTRI/2013/11/004133 (Registry Identifier: Clinical Trials Registry- India (CTRI))
Record Dates: First submitted 2018-03-09; First posted 2018-03-26 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Urinary Tract Infection Complicated; Acute Pyelonephritis
Keywords: CSE-1034 Double Blind Study; Elores; Meropenem; PLEA-CT; Bacterial Infections; ESBL; MBL; beta-lactamase; Anti-Infective Agents, Urinary; Anti-Infective Agents; Urinary Tract Infections; Pyelonephritis; Infection; Sulbactam; EDTA; Disodium EDTA; Antibiotic Adjuvant Entity; Antibiotic Resistance Breaker
MeSH Terms: conditions — Bacterial Infections; Urinary Tract Infections; Pyelonephritis; Infections | interventions — Ceftriaxone; Sulbactam; Edetic Acid; Meropenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSE-1034 (Ceftriaxone + Sulbactam + EDTA) (Experimental): CSE-1034 (Ceftriaxone + Sulbactam + EDTA) was an Experimental drug in this study and is a combination of Ceftriaxone 1000mg, Sulbactam 500mg and EDTA 37mg available as dry powder for reconstitution. It was administered twelve hourly through intravenous route as infusion over 30 minutes. The duration of the active treatment was for 5-14 days depending upon the severity of the disease, which was determined by the Principal Investigator (PI).
  Interventions:
  * Drug: CSE-1034 (Ceftriaxone + Sulbactam + EDTA)
  * Drug: Matching Placebo
  Interventions: Drug: CSE-1034 (Ceftriaxone + Sulbactam + EDTA)
- Meropenem (Active Comparator): Meropenem was the active comparator in the study. It was also available as dry powder for reconstitution and contained active ingredient Meropenem 1000mg. It was administered eight hourly through intravenous route as infusion over 30 minutes.The duration of the active treatment was for 5-14 days depending upon the severity of the disease, which was determined by the PI.
  Interventions:
  * Drug: Meropenem
  * Drug: Matching Placebo
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: CSE-1034 (Ceftriaxone + Sulbactam + EDTA) — CSE-1034 (Ceftriaxone + Sulbactam + EDTA) was Experimental in this study and is a combination of Ceftriaxone 1000mg, Sulbactam 500mg and EDTA 37mg available as dry powder for reconstitution. Patients were given either CSE-1034 or placebo through IV route four times daily, strictly adhering to the time interval. Time of the first dose (Drug) was considered 0th hr, the second dose (Placebo) was given at 8th hour from first dose, third dose (Drug) at 12th hour from first dose and the fourth dose (Placebo) at 16th hour from first dose. The infusion was initiated within ± 30 min of schedule time.
  Other Names: Elores
  Arms: CSE-1034 (Ceftriaxone + Sulbactam + EDTA)
Drug: Meropenem — Meropenem was the Comparator in the study. It was also available as dry powder for reconstitution and contained active ingredient Meropenem 1000mg.Patients were given either Meropenem or placebo through IV route four times daily, strictly adhering to the time interval. Time of the first dose (Drug) was considered 0th hr, the second dose (Drug) was given at 8th hour from first dose, third dose (Placebo) at 12th hour from first dose and the fourth dose (Drug) at 16th hour from first dose. The infusion was initiated within ± 30 min of schedule time.
  Other Names: Meronem
  Arms: Meropenem

SUMMARY:
The purpose of this study is to evaluate the effects of CSE-1034 (Ceftriaxone+ Sulbactam+ EDTA) compared to Meropenem for treating hospitalized patients with complicated urinary tract infections, including acute pyelonephritis caused by β-lactamase producing gram-negative bacteria

DETAILED DESCRIPTION:
cUTIs are mostly caused by gram-negative bacteria, including Enterobacteriaceae (particularly Escherichia coli, Klebsiella pneumoniae and Proteus mirabilis) and Pseudomonas aeruginosa, and often possess mechanisms leading to multidrug resistance. These mechanisms primarily consist of ESBLs (extended-spectrum beta-lactamases) that can hydrolyse cephalosporins, penicillins and aztreonam, and are encoded on mobile genes. This has led to increased risk of failure with first-line antibiotics and increased the usage of last line drugs like carbapenems. However, over the past decade, with the emergence of carbapenem-resistant infections caused by gram-negative pathogens like CRE (carbapenem-resistant Enterobacteriaceae), CRAB (carbapenem-resistant Acinetobacter baumannii) and CRPA (carbapenem-resistant Pseudomonas aeruginosa), there is a major threat looming on the effectiveness of these last resort drugs, warranting the discovery of newer and alternate agents.

To this end, the concept of using Antibiotic Resistance Breakers (ARBs) to revive the potency of existing antibiotics has been widely discussed in the recent literature. ARBs, sometimes referred as antibiotic adjuvants, are non-antibiotic moieties which do not have any antimicrobial activity on its own, but, in combination with antibiotics enhance their antimicrobial activity and help overcome resistance barriers. Most beta lactamase inhibitors (BLIs) can be thought of as ARBs that do not have any significant antimicrobial activity when used alone, but in combination with a beta-lactam antibiotic, help restore the activity against beta-lactamase producing organisms.

CSE-1034 is a novel combination of Ceftriaxone (third generation beta-lactam cephalosporin), Sulbactam (beta-lactamase inhibitor) and Disodium EDTA (Class 1 Antibiotic Resistance Breaker), and it restores the in vitro activity of Ceftriaxone against ESBL/MBL producing gram-negative bacteria, including enzyme families that belong to Ambler class A (TEM, SHV, CTX-M), class B (NDM, VIM, IMP), class C (some variants of AmpC), and class D (OXA ESBLs); it is not active against serine carbapenemases (higher variants of KPC, OXA carbapenemases). CSE-1034 also has proven in vitro activity against multiple resistance mechanisms including efflux pumps, bacterial biofilms, membrane permeability, and transfer of resistance by means of conjugation.

Since CSE-1034 has shown its efficacy in ESBL producing Escherichia coli, Klebsiella species, Pseudomonas aeruginosa and Acinetobacter species in various in vitro and in vivo studies, therefore, to meet regulatory expectations, non-inferiority of CSE-1034 in comparison to Meropenem (drug of choice in ESBL producing pathogens) is under study in this phase-3 clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing to provide informed consent and who are willing to or likely to comply with all study requirements
2. Patients of either gender must have age ≥ 18 years
3. Patients with suspected cUTI based on clinical signs and symptoms
4. Urine culture results confirm bacterial urinary tract infection caused by β-lactamase producing gram- negative bacteria requiring intravenous therapy
5. Patients with indwelling catheters should have the catheter removed or replaced (if removal is not clinically acceptable) before or as soon as possible, but not longer than 12 hours, after randomization
6. Obstructive uropathy, where the obstruction is likely to be relieved by stent or nephrostomy tube no later than 24 hours after randomization
7. Patients having received antibiotics for complicated urinary tract infection only if the duration of therapy was ≤ 24 hours within 72 hr of enrollment
8. Patients having received prior antibiotics and not showing any clinically significant improvement irrespective of duration of therapy
9. Females of childbearing potential require a negative urine pregnancy test and must agree to abstinence or to use an effective method of contraception

Exclusion Criteria:

1. Patients with clinically significant cardiovascular, renal, hepatic, gastrointestinal conditions, neurological, psychiatric, respiratory, other severely immunocompromised, haematological, or malignant disease and other condition which may interfere with the assessment. History of uncontrolled diabetes mellitus, HIV and hepatitis B were excluded.
2. Patients with history of resistance to any of the investigational drugs were excluded from the study
3. Patients with history of hypersensitivity or allergic response, any contra-indications to penicillin, cephalosporin groups of drugs
4. Patients with creatinine clearance below 30 mL/min
5. Patients having abnormal laboratory parameters which in the opinion of PI are clinically significant enough to pose any undue safety concern for the patient or can interfere with patient's assessment
6. Perinephritic abscess or renal corticomedullary abscess, polycystic kidney disease, only one functional kidney, chronic vesicoureteral reflux
7. Uncomplicated UTI
8. Previous or planned renal transplantation or cystectomy
9. Urinary tract surgery within 7 days prior to randomization or urinary tract surgery planned during the study period (except surgery to relieve obstruction, to place a stent or nephrostomy)
10. Patients with a Body Mass Index ≥ 35 kg/m^2
11. Pregnant or lactating women
12. Participation in any clinical study within the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2014-01-11 (Actual); Primary Completion 2017-05-08 (Actual); Study Completion 2017-05-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with symptomatic resolution (or return to premorbid state) of all UTI-specific symptoms (frequency/urgency/ flank pain / suprapubic pain) at the TOC visit in the Microbiological Modified Intent-To-Treat (mMITT) analysis set | TOC visit (16 to 25 days after randomization)
  This was the first co-primary outcome measure for the Food and Drug Administration (FDA). For this outcome measure, success was achieved with a clinical outcome of Cure at the Test of Cure (TOC) visit. Cure was defined as all or most pre-therapy signs and symptoms of the index infection had improved or resolved such that no additional antibiotics was required.
Proportion of patients with both a per-patient microbiological eradication and symptomatic resolution (or return to premorbid state) of all UTI-specific symptoms (frequency/urgency/ flank pain / suprapubic pain) at the TOC visit in the mMITT analysis set | TOC visit (16 to 25 days after randomization)
  This was the second co-primary outcome measure for the Food and Drug Administration (FDA). For this composite outcome measure, overall success was achieved with a clinical outcome of Cure and microbiologic outcome of Eradication at TOC visit. Cure was defined as all or most pre-therapy signs and symptoms of the index infection had improved or resolved such that no additional antibiotics was required. Eradication was defined using the FDA's colony-forming units per millilitre (CFU/mL) criteria that the bacterial pathogen(s) found at baseline was/were reduced to <10^4 CFU/mL of urine culture and a negative blood culture for an organism that was identified as an uropathogen (if repeated after positive at baseline blood culture).
Proportion of patients with a favorable per-patient microbiological response at the TOC visit in the mMITT analysis set | TOC visit (16 to 25 days after randomization)
  This was the primary outcome measure for the European Medicines Agency (EMA). For this measure, a microbiologic outcome of Eradication was defined using the EMA's CFU/mL criteria: bacterial pathogen(s) found at baseline was reduced to <10^3 CFU/mL of urine culture and a negative blood culture for an organism that was identified as an uropathogen (if repeated after positive at baseline blood culture).

SECONDARY OUTCOMES:
Proportion of patients with a favorable per-patient microbiological response in the mMITT analysis set | EOT (6 to 15 days after randomization) & LFU Visit (23 to 32 days after randomization)
  This secondary outcome measure focused on the microbiological success in the mMITT population at the End of Treatment (EOT), and Late Follow-Up (LFU) visits. A microbiologic outcome of Eradication was met if urine culture obtained at the relevant visit demonstrates <10^4 CFU/mL (for FDA) or < 10^3 CFU/mL (for EMA) of the original uro-pathogen, and the patient was not bacteremic (if the patient was bacteremic at Screening, the bacteremia has resolved)
Proportion of patients with a favorable per-patient microbiological response in the Microbiological Evaluable (ME) analysis set | EOT (6 to 15 days after randomization), TOC (16 to 25 days after randomization) & LFU Visit (23 to 32 days after randomization)
  This secondary outcome measure focused on the microbiological success in the ME population at the EOT, TOC, and LFU visits. A microbiologic outcome of Eradication was met if urine culture obtained at the relevant visit demonstrates <10^4 CFU/mL (for FDA) or < 10^3 CFU/mL (for EMA) of the original uro-pathogen, and the patient was not bacteremic (if the patient was bacteremic at Screening, the bacteremia has resolved)
Proportion of patients with a favorable per-patient microbiological response in the extended ME analysis set | EOT (6 to 15 days after randomization), TOC (16 to 25 days after randomization) & LFU Visit (23 to 32 days after randomization)
  This secondary outcome measure focused on the microbiological success in the extended ME population at the EOT, TOC, and LFU visits. A microbiologic outcome of Eradication was met if urine culture obtained at the relevant visit demonstrates <10^4 CFU/mL (for FDA) or < 10^3 CFU/mL (for EMA) of the original uro-pathogen, and the patient was not bacteremic (if the patient was bacteremic at Screening, the bacteremia has resolved)
Proportion of patients with symptomatic resolution (or return to premorbid state) of all UTI-specific symptoms (frequency/urgency/ flank pain / suprapubic pain) in the mMITT analysis set | EOT (6 to 15 days after randomization) & LFU Visit (23 to 32 days after randomization)
  This secondary outcome measure focused on a clinical outcome of Cure in the mMITT analysis set. For this outcome measure, success was achieved with a clinical outcome of Cure at the EOT, and LFU visit for mMITT population. Cure was defined as all or most pre-therapy signs and symptoms of the index infection had improved or resolved such that no additional antibiotics was required.
Proportion of patients with symptomatic resolution (or return to premorbid state) of all UTI-specific symptoms (frequency/urgency/ flank pain / suprapubic pain) in the CE analysis set | EOT (6 to 15 days after randomization), TOC (16 to 25 days after randomization) & LFU Visit (23 to 32 days after randomization)
  This secondary outcome measure focused on a clinical outcome of Cure in the Clinical Evaluable (CE) analysis sets. For this outcome measure, success was achieved with a clinical outcome of Cure at the EOT, TOC, and LFU visit for CE population. Cure was defined as all or most pre-therapy signs and symptoms of the index infection had improved or resolved such that no additional antibiotics was required.
Proportion of patients with symptomatic resolution (or return to premorbid state) of all UTI-specific symptoms (frequency/urgency/ flank pain / suprapubic pain) in the extended ME analysis set | EOT (6 to 15 days after randomization), TOC (16 to 25 days after randomization) & LFU Visit (23 to 32 days after randomization)
  This secondary outcome measure focused on a clinical outcome of Cure in the extended ME analysis set. For this outcome measure, success was achieved with a clinical outcome of Cure at the EOT, TOC, and LFU visit for extended ME population. Cure was defined as all or most pre-therapy signs and symptoms of the index infection had improved or resolved such that no additional antibiotics was required.
Proportion of favorable per-pathogen microbiological response in the mMITT analysis set | EOT (6 to 15 days after randomization), TOC (16 to 25 days after randomization) & LFU Visit (23 to 32 days after randomization)
  This secondary outcome measure focused on the per-pathogen (Enterobacter species, Escherichia coli, Proteus mirabilis, Pseudomonas aeruginosa and Acinetobacter baumannii) microbiological outcome of Eradication in the m-MITT population at EOT, TOC, and LFU visit. A microbiologic outcome of Eradication was met if urine culture obtained at the relevant visit demonstrates <10^4 CFU/mL (for FDA) or < 10^3 CFU/mL (for EMA) of the original uro-pathogen, and the patient was not bacteremic (if the patient was bacteremic at Screening, the bacteremia has resolved)
Proportion of favorable per-pathogen microbiological response in the ME analysis set | EOT (6 to 15 days after randomization), TOC (16 to 25 days after randomization) & LFU Visit (23 to 32 days after randomization)
  This secondary outcome measure focused on the per-pathogen (Enterobacter species, Escherichia coli, Proteus mirabilis, Pseudomonas aeruginosa and Acinetobacter baumannii) microbiological outcome of Eradication in the ME population at EOT, TOC, and LFU visit. A microbiologic outcome of Eradication was met if urine culture obtained at the relevant visit demonstrates <10^4 CFU/mL (for FDA) or < 10^3 CFU/mL (for EMA) of the original uro-pathogen, and the patient was not bacteremic (if the patient was bacteremic at Screening, the bacteremia has resolved)
Proportion of favorable per-pathogen microbiological response in the extended ME analysis set | EOT (6 to 15 days after randomization), TOC (16 to 25 days after randomization) & LFU Visit (23 to 32 days after randomization)
  This secondary outcome measure focused on the per-pathogen (Enterobacter species, Escherichia coli, Proteus mirabilis, Pseudomonas aeruginosa and Acinetobacter baumannii) microbiological outcome of Eradication in the extended ME population at EOT, TOC, and LFU visit. A microbiologic outcome of Eradication was met if urine culture obtained at the relevant visit demonstrates <10^4 CFU/mL (for FDA) or < 10^3 CFU/mL (for EMA) of the original uro-pathogen, and the patient was not bacteremic (if the patient was bacteremic at Screening, the bacteremia has resolved)
Proportion of patients with symptomatic resolution (as defined in the co-primary variables) for patients infected with a Meropenem -resistant pathogen in the extended ME analysis set | TOC visit (16 to 25 days after randomization)
  This secondary outcome measure focused on a clinical outcome of Cure in the patients infected with a Meropenem resistant pathogen in the extended ME analysis set. For this outcome measure, success was achieved with a clinical outcome of Cure at the TOC visit in extended ME population. Cure was defined as all or most pre-therapy signs and symptoms of the index infection had improved or resolved such that no additional antibiotics was required.
Proportion of patients with favorable per-patient microbiological response for patients infected with a Meropenem-resistant pathogen in the extended ME analysis sets | TOC visit (16 to 25 days after randomization)
  This secondary outcome measure focused on the microbiological success in the patients infected with a Meropenem-resistant pathogen in the extended ME analysis population at the TOC visit. A microbiologic outcome of Eradication was met if urine culture obtained at the relevant visit demonstrates <10^4 CFU/mL (for FDA) or < 10^3 CFU/mL (for EMA) of the original uro-pathogen, and the patient was not bacteremic (if the patient was bacteremic at Screening, the bacteremia has resolved)
Time to first defervescence while on IV study therapy in patients in the mMITT analysis set who had fever at study entry | EOT (6 to 15 days after randomization)
  This secondary outcome measure focused on the time to first defervescence in patients having fever study entry. Time to first defervescence was calculated for patients with a fever (>38°C) at Baseline. Defervescence (<37.8°C) was defined as absence of fever based on the highest temperature within a 24-hour period. Time to first defervescence while on IV study therapy (days) in the mMITT analysis set for patients who have fever at study entry was defined as the time from the first dose of IV study therapy to the first absence of fever.
Time to first defervescence while on IV study therapy in patients in the ME analysis set who had fever at study entry | EOT (6 to 15 days after randomization)
  This secondary outcome measure focused on the time to first defervescence in patients having fever study entry. Time to first defervescence was calculated for patients with a fever (>38°C) at Baseline. Defervescence (<37.8°C) was defined as absence of fever based on the highest temperature within a 24-hour period. Time to first defervescence while on IV study therapy (days) in the ME analysis set for patients who have fever at study entry was defined as the time from the first dose of IV study therapy to the first absence of fever.
Time to first defervescence while on IV study therapy in patients in the extended ME analysis set who had fever at study entry | EOT (6 to 15 days after randomization)
  This secondary outcome measure focused on the time to first defervescence in patients having fever study entry. Time to first defervescence was calculated for patients with a fever (>38°C) at Baseline. Defervescence (<37.8°C) was defined as absence of fever based on the highest temperature within a 24-hour period. Time to first defervescence while on IV study therapy (days) in the extended ME analysis set for patients who have fever at study entry was defined as the time from the first dose of IV study therapy to the first absence of fever.
Time to first defervescence while on IV study therapy in patients in the CE analysis set who had fever at study entry | EOT (6 to 15 days after randomization)
  This secondary outcome measure focused on the time to first defervescence in patients having fever study entry. Time to first defervescence was calculated for patients with a fever (>38°C) at Baseline. Defervescence (<37.8°C) was defined as absence of fever based on the highest temperature within a 24-hour period. Time to first defervescence while on IV study therapy (days) in the CE analysis set for patients who have fever at study entry was defined as the time from the first dose of IV study therapy to the first absence of fever.
Number of deaths due to cUTI with more than 5 days of treatment till TOC visit | EOT (6 to 15 days after randomization), TOC (16 to 25 days after randomization)
  This secondary outcome measure focused on the number deaths from day 01 dosing to TOC visit due to cUTI in patients received more than 5 days of treatment.
Total duration of treatment in the ME analysis sets | EOT (6 to 15 days after randomization)
  This secondary outcome measure focused on the number of days IV therapy was used for management of patients with cUTI including acute pyelonephritis
Total duration of treatment in the CE analysis sets | EOT (6 to 15 days after randomization)
  This secondary outcome measure focused on the number of days IV therapy was used for management of patients with cUTI including acute pyelonephritis
To measure the difference change in Patient Quality of life using Medical Outcome Study (MOS)-Short Form Survey (SF-36) scale | EOT (6 to 15 days after randomization), TOC (16 to 25 days after randomization) & LFU Visit (23 to 32 days after randomization)
  This secondary outcome measure focused on the MOS-SF-36 scale questionnaire. It was evaluated using the RAND methodology that measures the results based on eight different scales, namely - Physical functioning, Role limitations due to physical health, Role Limitations due to emotional problems, Energy/Fatigue, Emotional well-being, General Health, Health change, Pain and Social functioning. Broadly, the QoL scales are divided into two main sub-groups that provide a summary of the physical functioning and the mental functioning of the patient. Scores represent the percentage of the total possible score achieved, 100 being the highest score possible (denoting best outcome) and 0 being the lowest (denoting worst outcome)
Analysis of pharmacoeconomic data of CSE-1034 versus the comparator for mMITT population | EOT (6 to 15 days after randomization)
  This secondary outcome measure focused on Pharmacoeconomics data of CSE-1034 versus the Meropenem. The difference in cost incurred in management of cUTI (medications cost + hospitalization charges + cost of interventions and cost of laboratory investigations) were analyzed for mMITT population at EOT for CSE-1034 versus the comparator .
Analysis of pharmacoeconomic data of CSE-1034 versus the comparator for CE population | EOT (6 to 15 days after randomization)
  This secondary outcome measure focused on Pharmacoeconomics data of CSE-1034 versus the Meropenem. The difference in cost incurred in management of cUTI (medications cost + hospitalization charges + cost of interventions and cost of laboratory investigations) were analyzed for CE population at EOT for CSE-1034 versus the comparator .

OTHER OUTCOMES:
Safety endpoints-Incidence of Treatment Emergent Adverse Events (TEAE) in Safety Population | First infusion to Day 32
  Proportion of patients with any treatment-emergent adverse event reported during study period
Safety endpoints-Incidence of TEAE resulting in discontinuation of study drug therapy in Safety Population | From first infusion to last infusion of study therapy. Duration of study therapy was 1 to 14 days.
  Proportion of patients in the Safety analysis set for whom the assigned study treatment was discontinued, or interrupted.
Safety endpoints-Incidence of Serious Adverse Events (SAEs) in Safety Population | First infusion to Day 32
  Proportion of patients in the Safety analysis set who have any SAE during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev Sood, Principal Investigator — PGIMER Dr. RML Hospital, Baba Kharak Singh Marg, Connaught Place, New Delhi- 110001, India; Kim Mammen, Principal Investigator — Christian Medical College & Hospital, Ludhiana, Punjab-141008, India; R.P Agrawal, Principal Investigator — S.P. Medical College, Bikaner- 334003, Rajasthan, India; Manjunath M, Principal Investigator — Sapthagiri Institute of Medical Sciences and Research Center, #15, Chikkasandra, Hesaragatta Main Road, Bangalore-560 090, Karnataka, India; Pratibha Phadke, Principal Investigator — Deenanath Mangeshkar Hospital and Research Centre, Erandwane, Pune - 411004; Sudhir Chadha, Principal Investigator — Sir Ganga Ram Hospital, Rajinder Nagar, New Delhi- 110060, India; A.K. Deb, Principal Investigator — Sudbhawana Hospital, B 31/8023-B, Bhogabir, Lanka, Varanasi- 221005, India; Dharamraj Maurya, Principal Investigator — M.V. Hospital and Research Centre, 314/30, Mirza Mandi, Chowk, Lucknow- 226003, India; Deepak Dewan, Principal Investigator — Ajanta Hospital & Research Centre, 765, ABC Complex, Kanpur Road, Alambagh, Lucknow-Uttar Pradesh, 226005, India.; Shalini Srivastava, Principal Investigator — Om Surgical Centre and Maternity Home, SA 17/3, P-4, Sri Krishna Nagar, Paharia, Ghazipur Road, Varanasi- 221007, India; Ram Murti Singh, Principal Investigator — Trimurti Hospital, Gilat Bazaar, Varanasi- 221002, India; Rahul Janak Sinha, Principal Investigator — King George's Medical University (KGMU), Lucknow-226003, India; Madhav Prabhu, Principal Investigator — KLES, Dr Prabhakar Kore Hospital and Medical Centre, Nehru Nagar, Belagavi- 590010, Belgaum, Karnataka, India; Mohd. Shameem, Principal Investigator — J. N. Medical College, Aligarh Muslim University, Aligarh, Uttar Pradesh, India; Prem Nath Dogra, Principal Investigator — All India Institute of Medical Science, Ansari Nagar, New Delhi- 110029, India; Ravimohan S Mavuduru, Principal Investigator — P. G. I. M. E. R., Sector 12, Chandigarh-160012, India; Parvaiz Koul, Principal Investigator — SKIMS, Srinagar, Jammu & Kashmir- 190011, India
Locations (17):
- India (17):
  - Sher-i-Kashmir Institute of Medical Sciences (SKIMS), Srinagar, Jammu and Kashmir
  - Sapthagiri Institute of Medical Sciences and Research Center, Bangalore, Karnataka
  - KLES, Dr Prabhakar Kore Hospital and Medical Centre , , India, Belagavi, Karnataka
  - Deenanath Mangeshkar Hospital and Research Centre, Pune, Maharashtra
  - Christian Medical College & Hospital, Ludhiana, Punjab
  - S.P. Medical College, Bikaner, Rajasthan
  - J. N. Medical College, Aligarh Muslim University, Aligarh, Uttar Pradesh
  - King George's Medical University (KGMU), -, India, Lucknow, Uttar Pradesh
  - M.V. Hospital and Research Centre, Lucknow, Uttar Pradesh
  - Ajanta Hospital & Research Centre, 765, ABC Complex, Kanpur Road, Alambagh, -, , India., Lucknow, Uttar Pradesh
  - Trimurti Hospital, Varanasi, Uttar Pradesh
  - Sudbhawana Hospital, Varanasi, Uttar Pradesh
  - Om Surgical Centre and Maternity Home, Varanasi, Uttar Pradesh
  - P. G. I. M. E. R., Sector 12, - India, Chandigarh
  - PGIMER Dr. RML Hospital, New Delhi
  - All India Institute of Medical Science, New Delhi
  - Sir Ganga Ram Hospital, New Delhi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mir MDA, Chaudhary S, Payasi A, Sood R, Mavuduru RS, Shameem M. CSE (Ceftriaxone+ Sulbactam+ Disodium EDTA) Versus Meropenem for the Treatment of Complicated Urinary Tract Infections, Including Acute Pyelonephritis: PLEA, a Double-Blind, Randomized Noninferiority Trial. Open Forum Infect Dis. 2019 Oct 1;6(10):ofz373. doi: 10.1093/ofid/ofz373. PMID 31433059